CLINICAL TRIAL: NCT00623064
Title: Phase I Study of Cisplatin, Gemcitabine and Lapatinib as First Line Treatment in Advanced/Metastatic Urothelial Cancer
Brief Title: Lapatinib, Cisplatin, Gemcitabine as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-30061; EORTC-30061; EUDRACT-2006-002976-16; GSK-EORTC-30061
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: transitional cell carcinoma of the bladder; stage IV bladder cancer; stage III bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Lapatinib

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: lapatinib ditosylate
Other: pharmacological study

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib when given together with cisplatin and gemcitabine as first-line therapy in treating patients with locally advanced or metastatic urothelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended doses of lapatinib ditosylate when administered with gemcitabine hydrochloride and cisplatin, and determine on the basis of acute dose-limiting toxicity in course 1 in patients with locally advanced or metastatic transitional cell carcinoma of the urothelial tract.

Secondary

* To determine any relationship between drug exposure and adverse events in these patients.
* To assess the antitumor activity in these patients.

OUTLINE: This is a multicenter, dose-escalation study of lapatinib ditosylate.

* Lapatinib ditosylate, cisplatin, and gemcitabine hydrochloride: Patients receive oral lapatinib ditosylate once daily on days 1-28, cisplatin IV on day 2, and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity until the recommended dose of lapatinib ditosylate is determined.
* Lapatinib ditosylate, cisplatin, gemcitabine hydrochloride: Subsequently enrolled patients receive oral lapatinib ditosylate (beginning at one dose level below the recommended dose determined in the previous combination) once daily on days 1-21, cisplatin IV on day 1, gemcitabine hydrochloride IV over 30 minutes. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

All patients undergo blood sample collection periodically for pharmacokinetic analysis.

After completion of study treatment, patients are followed weekly.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven transitional cell carcinoma of the urothelial tract

  * Metastatic or locally advanced disease
* Measurable disease according to RECIST

  * Involvement of at least one target not in previously irradiated fields
* Overexpressing HER1 and/or HER2 receptors (HER2 3+ by IHC OR HER2 FISH or CISH positive)
* No clinical signs of CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* ANC ≥ 1,500/mm³
* Thrombocytes > 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 3 times ULN
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 3 months after completion of study treatment
* Cardiac ejection fraction normal
* Normal 12 lead ECG
* No serious cardiac illness or medical condition within the past 6 months including, but not limited to, any of the following:

  * Documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly controlled hypertension (e.g., systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg)
* No peripheral neuropathy > grade 1
* Able to swallow and retain oral medication
* No other malignancy within the past 3 years except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* No active or uncontrolled infections, serious illnesses, malabsorption syndrome or medical conditions, hepatitis, HIV, and/or cirrhosis
* No psychological, familial, sociological, or geographical condition potentially hampering study protocol compliance or follow-up schedule
* No current active hepatic or biliary disease (with the exception of Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver metastases or stable chronic liver disease)

PRIOR CONCURRENT THERAPY:

* Recovered from any effects of surgery
* Intravesicle therapy for superficial disease allowed
* Prior neoadjuvant or adjuvant chemotherapy allowed

  * Must have a minimum interval of six months between the completion of neoadjuvant or adjuvant chemotherapy and the diagnosis of metastatic disease
* No prior chemotherapy for metastatic disease
* No radiotherapy within the past 4 weeks
* No drugs and herbal inducers or inhibitors of CYP3A4 (e.g., bergamottin or glabridin) within 10 days prior to study treatment and while receiving lapatinib ditosylate therapy
* No other concurrent anticancer therapy or investigational agents
* No other concurrent anticancer agents
* No concurrent treatment with other investigational therapy for other diseases or conditions
* No concurrent prophylactic antibiotics
* No concurrent prophylactic filgrastim (G-CSF)
* At least 14 days since prior and no concurrent herbal or dietary supplements
* No concurrent consumption of grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lapatinib ditosylate in combination with cisplatin/gemcitabine hydrochloride and cisplatin/gemcitabine hydrochloride based on the documentation of the acute dose-limiting toxicity in course 1

SECONDARY OUTCOMES:
Pharmacokinetic profile of lapatinib ditosylate in combination with cisplatin/gemcitabine hydrochloride and cisplatin/gemcitabine hydrochloride
Antitumor activity according to RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark